CLINICAL TRIAL: NCT07239401
Title: Feasibility and Efficacy Trial of a Culturally Adapted Guided Self-Help CBT Manual for Obsessive-Compulsive Disorder: A Randomised Controlled Study From Pakistan
Brief Title: Feasibility and Efficacy Trial of a Culturally Adapted Guided Self-Help CBT Manual for OCD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Association of Cognitive Therapists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT_G_OCD_2025
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Obsessive - Compulsive Disorder
Keywords: OCD; Obsessive compulsive disorder; Guided self-help; CBT
MeSH Terms: conditions — Compulsive Personality Disorder; Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: This is a rater-blind, randomised controlled trial (RCT) comparing a guided self-help CBT intervention plus Treatment as Usual (TAU) with TAU alone. Participants will be randomly assigned (1:1 allocation) to either group. Assessments will occur at baseline and 12 weeks post-intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally adapted guided self-help OCD (Experimental): Participants will receive a culturally adapted guided self-help OCD manual based on culturally adapted CBT principles, designed to be used over ten weeks. The manual includes: Psychoeducation, Exposure and Response Prevention (ERP), Thought distraction techniques, Mood tracking and thought diaries, Identifying and modifying cognitive distortions, Problem-solving and communication strategies, and Relaxation and well-being exercises. Participants will receive the self-help manual at the time of initial assessment and intake, and then will be provided with telephone support. Psychology graduates working as guides will provide weekly telephone support. Intervention will be provided flexibly over 12 weeks. The second contact will be made at the time of final assessment on the 12th week.
  Interventions: Other: Culturally adapted Guided Self-Help OCD Manual
- Treatment as Usual (TAU) (No Intervention): Participants in the control group will receive standard outpatient care, which typically includes medication and brief consultation with psychiatrists or general practitioners. No formal psychological intervention will be offered during the study period. Pre-post assessment will be conducted over a 12-week span.

INTERVENTIONS:
Other: Culturally adapted Guided Self-Help OCD Manual — Participants will receive a culturally adapted guided self-help OCD manual based on culturally adapted CBT principles, designed to be used over ten weeks. The manual includes: Psychoeducation, Exposure and Response Prevention (ERP), Thought distraction techniques, Mood tracking and thought diaries, Identifying and modifying cognitive distortions, Problem-solving and communication strategies, and Relaxation and well-being exercises. Participants will receive the self-help manual at the time of initial assessment and intake, and then will be provided with telephone support. Psychology graduates working as guides will provide weekly telephone support. Intervention will be provided flexibly over 12 weeks. The second contact will be made at the time of final assessment on the 12th week.
  Arms: Culturally adapted guided self-help OCD

SUMMARY:
This randomised controlled trial (RCT) aims to assess the feasibility, acceptability, and preliminary efficacy of a culturally adapted, guided self-help cognitive behaviour therapy (CBT) manual specifically designed for individuals with OCD in Pakistan.

DETAILED DESCRIPTION:
Obsessive-Compulsive Disorder (OCD) is a chronic and debilitating mental health condition characterised by persistent, intrusive thoughts (obsessions) and repetitive behaviours or mental acts (compulsions). These symptoms are often distressing, time-consuming, and cause significant functional impairment and reduction in quality of life. Cognitive and behavioural therapies, particularly the Exposure and Response Prevention (ERP), have consistently demonstrated efficacy as a first-line treatment for OCD. However, access to trained therapists remains limited in low- and middle-income countries (LMICs), including Pakistan.

Self-help interventions rooted in CBT principles, especially when culturally adapted, represent a promising, scalable, and cost-effective alternative to conventional therapy. Previous research in Pakistan has shown the feasibility and acceptability of culturally adapted CBT (CaCBT) in treating depression and OCD within primary care and outpatient settings (Naeem et al., 2011; Aslam et al., 2015).

This randomised controlled trial (RCT) aims to assess the feasibility, acceptability, and preliminary efficacy of a culturally adapted, guided self-help CBT manual specifically designed for individuals with OCD in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical diagnosis of OCD (with or without comorbid depression)
* Minimum 5 years of formal education
* Residing within commuting distance of the participating sites
* Ability to read and write Urdu
* Provision of informed written consent

Exclusion Criteria:

* Current substance use or dependence (diagnosed)
* Significant cognitive impairment (e.g., dementia or intellectual disability)
* OCD with active psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Obsessive-compulsive symptoms | 12 weeks
  As assessed through participants' scores on the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS)
Feasibility and acceptability | 12 weeks
  Feasibility and acceptability will be assessed through trial procedure, recruitment, retention and informal feedback from participants.
Clients' satisfaction | 12 weeks
  The client satisfaction scale will be used. At the end of the intervention, researchers will ask participants to describe their experience. They will be asked to name the sessions they found most or least helpful and to provide suggestions for improving the intervention.

SECONDARY OUTCOMES:
Anxiety & depression | 12 weeks
  As assessed through participants' scores on the Hospital Anxiety and Depression Scale (HADS)
Functionality | 12 weeks
  As assessed through participants' scores on the WHO Disability Assessment Schedule 2 (WHODAS 2)

CONTACTS AND LOCATIONS:
Overall Officials: Mirrat Gul Butt, PhD, Principal Investigator — Pakistan Association of Cognitive Therapists

IPD SHARING:
Plan to Share IPD: No